CLINICAL TRIAL: NCT03331718
Title: PoLyglycolic Acid Felt reiNforcEmenT of the PancreaticoJejunostomy; Multicenter Prospective Randomized Phase III Trial in Japan and Korea (PLANET-PJ Trial)
Brief Title: PoLyglycolic Acid Felt reiNforcEmenT of the PancreaticoJejunostomy (PLANET-PJ Trial)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toyama (Other)
Collaborators: Seoul National University Hospital (Other); Kansai Medical University (Other); Kumamoto University (Other); Nagoya University (Other); Nara Medical University (Other); Osaka City University (Other); Osaka University (Other); Shiga Medical University (Unknown); Shimane University (Unknown); Tokyo Medical and Dental University (Other); Tokyo Medical University (Other); Wakayama Medical University (Other); Gangnam Severance Hospital (Other); National Cancer Center, Korea (Other Government); Samsung Medical Center (Other); Seoul National University Bundang Hospital (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Tsutomu Fujii, MD, PhD, FACS, University of Toyama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PLANET-PJ
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Disease of Pancreatic or Periampullary Lesions
Keywords: pancreatoduodenectomy; pancreaticojejunostomy; polyglycolic acid; Neoveil; pancreatic fistula; pancreas
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Pancreaticojejunostomy with duct-to-mucosa anastomosis is performed as usual.
- PGA felt reinforcement (Active Comparator): In addition to usual pancreaticojejunostomy, PGA felt is used in duplicate.
  Interventions: Drug: PGA felt reinforcement

INTERVENTIONS:
Drug: PGA felt reinforcement — During pancreaticojejunostomy, 1) a 0.3 mm thick PGA felt (Neoveil®, Gunze, Japan) is pasted on the ventral side and the dorsal side of pancreatic parenchyma, through which suture between pancreatic parenchyma and jejunum is performed. 2) Before abdominal closure (after completion of all reconstruction, after washing in the abdominal cavity), a 0.15 mm thick PGA felt is further covered around the anastomotic site and fibrin glue is sprayed.
  Arms: PGA felt reinforcement

SUMMARY:
The polyglycolic acid (PGA) felt is a felt-like absorbable suture reinforcing material. The pancreatojejunostomy aimed at reducing POPF is not established at present. We devised a new method using doubly PGA felt. This study is a multicenter, randomized phase III trial between Japan and Korea to verify the usefulness of this double coating of PGA felt.

DETAILED DESCRIPTION:
Pancreatojejunostomy is generally a combination of suture between the pancreatic parenchyma and the seromuscular layer of the jejunum, and duct-to-mucosa suture. The clinical study about the various kinds of pancreatojejunostomy have been reported for the purpose of lowering the frequency of POPF; however, the frequency of more than grade B POPF is still around 10 to 20%. In soft pancreas cases with unexpanded pancreatic ducts, the risk is further elevated.

The polyglycolic acid (PGA) felt is an absorbable suture reinforcing material. It is generally used to reinforce sutures of fragile tissues such as the lung, bronchi, liver, and gastrointestinal tract, and to reinforce a wide range of tissue defects. Regarding pancreatojejunostomy using a PGA felt, the incidence of POPF formation was decreased in some retrospective studies; on the other hand, no significant difference was found in other study. As described above, the pancreatojejunostomy aimed at reducing POPF is not established at present. We devised a new method using doubly PGA felt. This study is a multicenter, randomized phase III trial between Japan and Korea to verify the usefulness of this double coating of PGA felt.

ELIGIBILITY:
Inclusion Criteria:

1. Disease of pancreatic or periampullary lesions to require pancreatoduodenectomy
2. Planned pancreaticojejunostomy including duct-to-mucosa anastomosis
3. MPD diameter ≤3mm on the left side of the portal vein in preoperative imaging (CT or MRI)
4. Performance status (ECOG scale): 0-1 at the time of enrollment
5. Age: 20 years or older
6. Adequate organ function A) Leukocyte count: ≥2500 mm3, ≤14000 mm3 B) Hemoglobin: ≥9.0 g/dL C) Platelet count: ≥100,000 mm3 D) Total Bilirubin: ≤2.0 mg/dL (not apply to cases with obstructive jaundice) E) Creatinine: ≤2.0 mg/dL
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Planned pancreatogastrostomy
2. Laparoscopic or laparoscope-assisted pancreatoduodenectomy
3. Pancreatic parenchymal atrophy or calcification due to chronic pancreatitis
4. Neoadjuvant treatment including chemotherapy or radiotherapy
5. History of upper abdominal surgery (both of open and laparoscopic) except cholecystectomy
6. Emergency operation
7. Arterial reconstruction such as superior mesenteric artery, common hepatic artery, or celiac artery
8. Severe ischemic heart disease
9. Severe liver dysfunction due to liver cirrhosis or active hepatitis
10. Severe respiratory disorder required oxygen inhalation
11. Chronic renal failure with dialysis
12. Requiring resection of other organs (liver or colon) during pancreatoduodenectomy
13. Immunosuppressive treatment
14. History of severe hypersensitivity to PGA felt and fibrin glue
15. Other severe drug allergies
16. Contrast media allergy of both iodine and gadolinium
17. Active duplicate cancer thought to affect adverse events
18. Severe psychological or neurological disease
19. Drug abuse or alcoholics
20. Planned use of octreotide

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of a clinically relevant POPF (ISGPS grade B/C) | within 3 months after surgery
  Incidence of a clinically relevant POPF (grade B/C), according to the ISGPS criteria which is the evaluation criteria for POPF

SECONDARY OUTCOMES:
Length of drain placement | within 3 months after surgery
  Number of days from operation date to drain removal date (the peripancreatic drain to be removed last)
Length of the hospital stay | within 3 months after surgery
  Number of days from operation date to discharge date
Incidence of overall POPF (Biochemical leak, grade B, and C) | within 3 months after surgery
  Incidence of overall POPF of biochemical leak, grade B, or grade C, according to the ISGPS criteria
Incidence of POPF by each suturing method to approximate the pancreas and the jejunum | within 3 months after surgery
  Incidence of overall POPF of biochemical leak, grade B, or grade C, according to the ISGPS criteria by each suturing method to approximate the pancreas and the jejunum (Kakita, two-layer, or Blumgart)
Incidence of delayed gastric emptying (DGE) | within 3 months after surgery
  Incidence of overall DGE, according to the ISGPS criteria
Incidence of intraabdominal abscess | within 3 months after surgery
  Incidence of intraabdominal abscess of Grade II (requiring pharmacological treatment with drugs) or more, according to Clavien-Dindo classification
Incidence of postpancreatectomy hemorrhage (PPH) | within 3 months after surgery
  Incidence of overall PPH, according to the ISGPS criteria
Incidence of interventional drainage | within 3 months after surgery
  Incidence of additional drainage percutaneously or endoscopically
Incidence of overall postoperative complications | within 3 months after surgery
  Incidence of overall postoperative complications, according to Clavien-Dindo classification
Incidence of POPF-related complications (POPF+DGE+abscess+PPH) | within 3 months after surgery
  Incidence of cases in whom one of 3), 5), 6) or 7) occurred
Incidence of 3-month mortality | within 3 months after surgery
  Incidence of surgery-related deaths from operation date to postoperative 3 months
Incidence of reoperation | within 3 months after surgery
  Incidence of reoperation from operation date to postoperative 3 months
Incidence of readmission | within 3 months after surgery
  Incidence of readmission from operation date to postoperative 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Fujii, MD, PhD, Principal Investigator — University of Toyama
Locations (1):
- University of Toyama, Toyama, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shibuya K, Park JS, Kwon W, Kawai M, Yoshioka I, Hashimoto D, Takami H, Lim CS, Seo HI, Nagai M, Inoue Y, Yoon YS, Lee SE, Baba H, Choi SB, Lee HK, Do Yang J, Kimura Y, Hwang HK, Nah YW, Tani M, Akahoshi K, Han IW, Nagakawa Y, Eguchi H, Yamada S, Satoi S, Sho M, Kitayama M, Wan K, Shimokawa T, Yamaue H, Jang JY, Fujii T. Effect of Double Layer Polyglycolic Acid Felt for Reducing Pancreatic Fistula After Pancreatoduodenectomy: Results of a Multicenter Randomized Control Trial (PLANET-PJ trial). Ann Surg. 2025 Jul 29. doi: 10.1097/SLA.0000000000006857. Online ahead of print. PMID 40728222
- [Derived] Shibuya K, Jang JY, Satoi S, Sho M, Yamada S, Kawai M, Kim H, Kim SC, Heo JS, Yoon YS, Park JS, Hwang HK, Yoshioka I, Shimokawa T, Yamaue H, Fujii T. The efficacy of polyglycolic acid felt reinforcement in preventing postoperative pancreatic fistula after pancreaticojejunostomy in patients with main pancreatic duct less than 3 mm in diameter and soft pancreas undergoing pancreatoduodenectomy (PLANET-PJ trial): study protocol for a multicentre randomized phase III trial in Japan and Korea. Trials. 2019 Aug 9;20(1):490. doi: 10.1186/s13063-019-3595-x. PMID 31399139